CLINICAL TRIAL: NCT02951923
Title: The Effect of 8-weeks of Bovine Colostrum and Soy Protein Supplementation on Fitness, Muscle Mass, Inflammation and Immune Function During Intense Training in Rugby Players
Brief Title: The Effect of 8-weeks of Bovine Colostrum and Soy Protein Supplementation in Rugby Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Ph.D., University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIO14-81
Record Dates: First submitted 2014-12-01; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Exercise Performance; Body Composition

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bovine colostrum (Experimental): 8 weeks of Bovine colostrum power, 60g per day
  Interventions: Dietary Supplement: Bovine Colostrum
- Soy powder (Active Comparator): 8 weeks of Soy powder, 60g per day
  Interventions: Dietary Supplement: Soy

INTERVENTIONS:
Dietary Supplement: Bovine Colostrum — Bovine colostrum vs. soy during rugby training
  Arms: Bovine colostrum
Dietary Supplement: Soy
  Arms: Soy powder

SUMMARY:
Bovine colostrum is the milk produced by cows immediately after calving. It contains high levels of proteins that improve immune protection and may act to prevent colds. During intense training, athletes often have compromised immune function. This may be especially true in club-level rugby players who abruptly start high intensity training in the spring in preparation for their competitive season. Our study will assess the effects of supplementing these players with bovine colostrum during this intense training. Thirty-six players will be recruited; half will consume colostrum during the 8 weeks of early-season training and half soy protein. The investigators predict the bovine colostrum supplement will improve health during the training and increase fitness levels.

DETAILED DESCRIPTION:
Bovine colostrum is the first milk secreted by cows after calving. Colostrum is high in protein and contains a number of bioactive substances including growth and antimicrobial factors. Antimicrobial factors in bovine colostrum include immunoglobulin and a variety of other less specific antimicrobial proteins and peptides. Immunoglobulin and other antimicrobials are important for immune system function. This is important to athletes because intense exercise training can compromise the immune system; therefore bovine colostrum has potential to improve exercise performance by preventing immune system dysfunction that is common during periods of heavy exercise training .

Preliminary studies of colostrum supplementation show its potential for increasing human exercise performance. The mechanism through which colostrum acts to benefit performance remains unclear. Similarly, further studies are required to elucidate colostrum-induced effects in individuals of different ages and levels/intensity of physical activity.

The main growth factor in bovine colostrum is insulin-like growth factor-1 (IGF-1). Bovine colostrum supplementation in young individuals increased IGF-1 levels. Insulin-like growth factor-1 stimulates growth of muscle tissue and is important in maintaining muscle mass and function in adults.

Bovine colostrum supplementation has been shown to increase lean tissue (muscle mass) in younger individuals. Eight to 12 weeks of bovine colostrum supplementation during a resistance training program increased lean tissue mass by 1.5 to 2 kg compared to increases of 0 to 1.2 kg while on whey protein supplementation. We have also recently shown that bovine colostrum supplementation increases muscular strength compared to similar amounts of supplementation with whey protein in men and women over 50y.

Examining the effects of colostrum in rugby players presents a unique scientific opportunity because of the nature of their training regime. Rugby players' early season workouts are the most stressful training sessions of the season (after the winter break they must condition quickly for the start of the season with few if any pre-season games and their workouts involve repeated sprint activity in addition to weight training). Rugby players would be most susceptible to overtraining and immune system depression during this time of the year. Bovine colostrum with its high levels of anti-microbials and other bioactive factors may be beneficial to mitigate the deleterious effects of early, high intensity training.

The objective of the proposed internship study is to determine the effects of 8 weeks of bovine colostrum supplementation, compared to soy protein supplementation in rugby players during early season training.

ELIGIBILITY:
Inclusion Criteria:

* active rugby players

Exclusion Criteria:

* Not taking nutritional supplements within one month of the study
* Answered "yes" to a physical activity readiness questionnaire indicating health problems that could be exacerbated with physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in lean tissue mass | baseline, 8 weeks
Change in leg press strength | baseline, 8 weeks
Change in bench press strength | baseline, 8 weeks
Change in aerobic capacity as predicted by the Leger shuttle run test | baseline, 8 weeks
Change in leg power as assessed by vertical jump height | baseline, 8 weeks

SECONDARY OUTCOMES:
Change in salivary immunoglobulin A | baseline, 8 weeks
Change in salivary interleukin 6 | baseline, 8 weeks
Change in salivary interleukin 1-beta | baseline, 8 weeks
Change in salivary c-reactive protein | baseline, 8 weeks
Incidence of upper respiratory tract infections | Up to 8 weeks
Adverse events | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chilibeck, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- College of Kinesiology, University of Saskatchewan, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Duff WR, Chilibeck PD, Rooke JJ, Kaviani M, Krentz JR, Haines DM. The effect of bovine colostrum supplementation in older adults during resistance training. Int J Sport Nutr Exerc Metab. 2014 Jun;24(3):276-85. doi: 10.1123/ijsnem.2013-0182. Epub 2013 Nov 25. PMID 24281841